CLINICAL TRIAL: NCT05155618
Title: Intervention Study on Life Style and Microbiota in Prostate Cancer Patients Undergoing Radiotherapy
Brief Title: Intervention Study in Prostate Cancer Patients Undergoing Radiotherapy
Acronym: MicroStyle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Collaborators: Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IEO 1442
Record Dates: First submitted 2021-09-14; First posted 2021-12-13 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2023-06

CONDITIONS: Prostate Cancer
Keywords: Lifestyle; microbiota; diet; radiotherapy; physical activity
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Supportive Care: protocol designed to evaluate one or more interventions where the primary intent is to maximize comfort, minimize side effects or mitigate against a decline in the subject's health or function. In general, supportive care interventions are not intended to cure a disease.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (IG) (Experimental): Participants randomized to the IG will be offered an individualized counseling during cancer treatments that includes both a dietary and physical activity suggestions to control side effects, to cope with feelings of anxiety or depression and to improve quality of life.
  Interventions: Procedure: INTERVENTION GROUP
- Control group (CG) (No Intervention): Participants included in the CG will receive at baseline general advice and materials available for patients undergoing RT. According to the crossover design, the CG will cross to the intervention as proposed for the IG, after the initial 6-month period.

INTERVENTIONS:
Procedure: INTERVENTION GROUP — Personalized advice to prevent side effect according to their health status will be provided by a dietitian and a physiotherapist.
  Other Names: IG
  Arms: Intervention group (IG)

SUMMARY:
Microstyle study aims to evaluate the effect of a 6-month intervention in a group of prostate cancer patients undergoing radiotherapy. Intervention is designed to control side effects and to improve adherence to a healthy lifestyle (diet and increase level of physical activity and decreased sedentary time) measured by the change in adherence to a healthy lifestyle score. The impact of the intervention on toxicity and gastrointestinal symptomatology will be measured by a mediation framework analysis. This approach allows investigating how microbiome may mediate effect of treatment. It will be also assessed the change in microbiome in relation to the change in cytokines/ adipokines in association with early and late toxicity.

DETAILED DESCRIPTION:
MicroStyle study is a randomized two-arm crossover clinical trial. Study participants will be recruited among men undergoing radiotherapy (RT) in two centers (Milan and Naples). The study will be conducted over a three-year period, during which patients will receive a 6-month intervention and will be followed for other 6 months. The crossover design is used to reduce drop-out and to offer all patients the same opportunities, and also to evaluate the effect of the intervention after 6-month from RT when patients should have recreated a healthier microbiome and have less treatment side effects.

Three hundred patients will be enrolled over the study period and randomized in two arms: Intervention Group (IG) and Control Group (CG). Participants allocated to the IG will meet a dietitian and a physiotherapist before RT to receive personalized diet and exercise recommendations, according to their health status, to improve overall lifestyle and reduce side effects (bowel and/or urinary problems). The dietitian will give indication to limit the gastrointestinal side effects reducing consumption of foods rich in fiber, lactose and simple sugars, and the physiotherapist will set individualized goals based on capabilities, lifestyle pattern and preferences to increase physical activity and to reduce sedentary time. Moreover, the physiotherapist will provide specific indication to improve genitourinary health to reduce urinary incontinence that follows prostate treatments, erectile dysfunction and pelvic pain due to muscle spasm. All participants will be given a pedometer device (steps counter) in order to monitor and interfere (in the intervention group) with participants' physical activity and sedentary time. Participants included in the CG will receive at baseline general advice and materials available for patients undergoing RT. According to the crossover design, the CG will cross to the intervention as proposed for the IG, after the initial 6 months period.

Microstyle study foresee a 6-month intervention followed by 6-months of follow-up, over a period of 12 months for the intervention group (IG) while the control group (CG) will start the intervention 6 months after RT and they will follow-up for other 6 months over a period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* men aged 18 or older
* candidates for a prostate curative treatment with RT (which includes exclusive RT +/-hormone therapy, surgery followed by RT +/- hormone therapy) AND
* good performance status (ECOG < 2) AND
* written informed consent obtained AND
* willing to be randomized to either group, AND
* willing to wear the wrist-based activity monitor during the 6-month study period.

Exclusion Criteria:

* BMI <18.5 AND
* extra pelvic lymph node involvement or metastasis and severe medical condition(s) that would prevent optimal participation in the physical activities prescribed AND
* Malnutrition Universal Screening Tool (MUST) ≥ 2. It considers body mass index, weight change and acute disease effect equally and determines a malnutrition risk score. A score ≥2 identify a patient at high risk of malnutrition AND
* investigator does not approve participation in the study in case of severe clinical condition that would prevent optimal participation in the physical activities prescribed; any other severe medical condition or advanced age impeding the patient to adhere at the planned study follow-up period.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in adherence to a healthy lifestyle score | It will be assessed at the end of the 6-month intervention
  The score will be computed using BMI, level of physical activity and food consumptions according the standardized system based on the World Cancer Research Fund (WCRF) and the American Institute for Cancer Research (AICR) recommendations (Shams-White et al, 2019). The score will range from 0 (minimal adherence) to 7 (maximal adherence).

SECONDARY OUTCOMES:
The effects of the interventions on serum biomarkers | 6-month - 12-month and 18-month (only for the CG)
  differences by arms in changes of Prostate-specific antigen (PSA) (mcg/L) and 25-hydroxyvitamin D (ng/mL) compared to the baseline.
Change in body composition | 6-month - up to 30 days - 12-month and 18-month (only for the CG)
  change in body composition assessed at all visits using bioelectrical impedance vector analysis (BIVA) compared to the baseline
Change in quality of Life | 6-month - 12-month and 18-month (only for the CG)
  change in quality of life, measured by the Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire which consists of 39 items. Each item is rated on a 0 to 4 Likert type scale, and then combined to produce subscale scores. Higher scores represent better QoL.
Change in Dietary intake | 6-month - up to 30 days - 12-month and 18-month (only for the CG)
  change in daily or weekly intake of the main food groups included in a validated short self-administered questionnaire over the previous months and the change over the study
change in the level of physical activity | 6-month and 12-month (only for the CG)
  The International Physical Activity Questionnaire (IPAQ)- Short Form will be used. It obtains information about how much time is spent while walking and in moderate and vigorous activities and sitting duration in the last 7 days. The questionnaire records the activity of four intensity levels: 1) vigorous-intensity activity, 2) moderate-intensity activity, 3) walking, and 4) sitting. Durations are multiplied by known metabolic equivalent of tasks (METs) per activity and the results for all items are summed for the overall physical activity score. Scores for walking and for moderate and vigorous activities are sums of corresponding item scores. The change in the level of physical activity will be estimated and compared to the baseline.
Change in acute and late toxicity | 6-month - up to 30 days - 12-month and 18-month (only for the CG)
  change in toxicity according to Radiation Therapy Oncology Group/European Organisation for Research and Treatment of Cancer (RTOG/EORTC) scoring criteria. It consists of a scoring range from 0 to 5 where 0 means an absence of radiation effects and 5 means the effects led to death, compared to the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Gandini, MSc, Principal Investigator — Department of Experimental Oncology, IEO, Milan; Valentina Borzillo, MD, Principal Investigator — Department of Radiation Oncology, Istituto Nazionale Tumori IRCCS Fondazione G Pascale, Napoli
Locations (2):
- Italy (2):
  - European Institute of Oncology, Milan
  - Istituto Nazionale Tumori-IRCCS-Fondazione G. Pascale, Naples

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gnagnarella P, Marvaso G, Jereczek-Fossa BA, de Cobelli O, Simoncini MC, Nevola Teixeira LF, Sabbatini A, Pravettoni G, Johansson H, Nezi L, Muto P, Borzillo V, Celentano E, Crispo A, Pinto M, Cavalcanti E, Gandini S; MicroStyle Collaborative Group. Life style and interaction with microbiota in prostate cancer patients undergoing radiotherapy: study protocol for a randomized controlled trial. BMC Cancer. 2022 Jul 19;22(1):794. doi: 10.1186/s12885-022-09521-4. PMID 35854230